CLINICAL TRIAL: NCT07123038
Title: A Long-Term Follow-Up Observational Study to Evaluate Safety in Subjects Who Have Received a Gene-Modified Regulatory T Cell (Treg) Therapeutic
Status: Recruiting | Type: Observational
Sponsor: Sonoma Biotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SBT0000-01
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis (RA); Hidradenitis Suppurativa (HS)
Keywords: Rheumatoid Arthritis; Long Term Follow Up Study; Treg; SBT0000-01; Hidradenitis Suppurativa; SBT777101; SBT777101-01; SBT777101-02
MeSH Terms: conditions — Arthritis, Rheumatoid; Hidradenitis Suppurativa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants exposed to SBT777101 Treg cell therapy: Participants exposed to SBT777101 during the original Phase 1 clinical safety study (NCT06201416, NCT06361836)
  Interventions: Other: Long Term Safety Monitoring Procedures

INTERVENTIONS:
Other: Long Term Safety Monitoring Procedures — In accordance with the schedule of assessments, participants will complete the long term safety and health questionnaire and will undergo routine physical examinations. A review will be conducted on selected adverse events, medical history, and concomitant medication use. Collection of biospecimens (blood and tissue) will be taken as appropriate at scheduled visits to monitor for delayed adverse events related to prior cell therapy.

SUMMARY:
To assess the emergence, type, severity, and potential causality of delayed adverse events following administration of a gene-modified Treg therapeutic.

DETAILED DESCRIPTION:
The purpose of this LTFU study is to evaluate safety (delayed adverse events) for up to 15 years in subjects who have received a gene-modified Treg therapeutic within clinical studies NCT06201416, NCT6361836. This is a Phase 4, multi-center long-term follow-up observational study to evaluate long-term safety in subjects who have received a gene-modified Treg therapeutic across Sonoma Biotherapeutics, Inc. clinical studies. The duration of the study is up to 15 years after dose of a Treg therapeutic in prior parent treatment protocols (SBT777101-01 and SBT777101-02) conducted by the Sponsor. Study visits will occur in accordance with the Schedule of Assessments.

ELIGIBILITY:
Inclusion Criteria:

* Subject was previously administered at least 1 dose of a Sonoma Biotherapeutics, Inc. gene-modified Treg therapeutic in a prior parent treatment protocol.
* Subject understands the purpose and risks of the study and is willing to provide written informed consent.
* Subject is willing to comply with all study procedures for the follow-up period.

Exclusion Criteria:

* Participation in the study is not in the subject's best interest, in the opinion of the Investigator

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrolled participants will be determined by the number of subjects participating in the SBT777101-01 and SBT777101-02 studies.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-07-22 (Actual); Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of delayed adverse events considered at least possibly related to the SBT777101 gene-modified Treg therapeutic | 15 years

SECONDARY OUTCOMES:
Persistence of the SBT777101 gene-modified Treg therapeutic | 15 years
Incidence of replication competent lentivirus (RCL) | 15 years
Mortality in patients who received a gene-modified Treg therapeutic | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mei-Lun Wang, MD, Study Director — Sonoma Biotherapeutics
Locations (10):
- United States (10):
  - UCSF Medical Center, San Francisco, California
  - Stanford Medical Center, Stanford, California
  - University of Colorado, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Tufts University, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Duke University, Durham, North Carolina
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No